CLINICAL TRIAL: NCT06564220
Title: Testicular Adrenal Rest Tumor in Congenital Adrenal Hyperplasia Patients Attending Assiut University Children Hospital
Brief Title: Testicular Adrenal Rest Tumor in Congenital Adrenal Hyperplasia Patients Attending Assuit University Children Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Refaat Zain El-Abidin Zahran, 71515,Assuit, Assiut University
Other Study IDs: Testicular adrenal rest tumor
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Testicular Adrenal Rest Tumor; Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
assessment of the risk factors contributing for TART development in a male child with congenital adrenal hyperplasia.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is one of the most frequent endocrine disorders. It is characterized by deficient activity of one of the enzymes necessary for adrenal Cortisol synthesis. Autosomal recessive inheritance of deficient 21-hydroxylase (21 OH) activity accounts for more than 90% of cases. [1]

One of the most important and frequently detected complications in males with congenital adrenal hyperplasia (CAH) is the development of testicular adrenal rest tumours (TARTs). . [2],[3]

Testicular adrenal rest tumor is a benign tumor originating from adrenal cells within the testicles; the adrenal cells migrate at 8 weeks of gestation from the urogenital ridge along with the gonadal cells to the testicle. The exact mechanism underlying tumor growth and development is still not well understood . [4],[5]

The correct diagnosis of TART is important for differential diagnosis with malignant testis tumors, which need orchiectomy, as opposed to TART, usually treated exclusively with exogenous steroids. [6].

Although TARTs are always benign, their location in the rete testis could obstructs the seminiferous tubules and causes gonadal dysfunction and infertility. Therefore, it is important to detect and treat TARTs at an early stage, especially in adolescents or young adults. [5],[7]

testicular ultrasound should be done in order to evaluate the presence of these lesions, its size, location, and characteristics. [9]

TARTs in children have mostly been presented as case reports in the literature, and only a limited number of studies have described the prevalence of TARTs in large populations of children . [2],[8]

As not all male CAH patients are affected by this complication, attempts have been made to identify the risk factors for the development of TARTs . [7]

ELIGIBILITY:
Inclusion Criteria:

* All male patients diagnosed as congenital adrenal hyperplasia based on clinical manifestations and laboratory investigations from age of 4 years to age of 18 years.

Exclusion Criteria:

* Patients with other adrenal insufficiency cause and Congenital adrenal hyperplasia that progressed to true precocious puberty

Ages: 4 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes
Study Population: male patients diagnosed as congenital adrenal hyperplasia based on clinical manifestations and laboratory investigations from age of 4 years to age of 18 years.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Testicular adrenal rest tumor in congenital adrenal hyperplasia patients attending Assiut University Children Hospital | Baseline
  Assessment of risk factors contributing for TART development in a child with congenital adrenal hyperplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa K Mohamed, Study Director — Lecturer of pediatric, faculty of medicine Assiut University

REFERENCES:
- [Background] Grunieiro-Papendieck L, Chiesa A, Mendez V, Prieto L. Neonatal screening for congenital adrenal hyperplasia: experience and results in Argentina. J Pediatr Endocrinol Metab. 2008 Jan;21(1):73-8. doi: 10.1515/jpem.2008.21.1.73. PMID 18404975
- [Background] Aycan Z, Bas VN, Cetinkaya S, Yilmaz Agladioglu S, Tiryaki T. Prevalence and long-term follow-up outcomes of testicular adrenal rest tumours in children and adolescent males with congenital adrenal hyperplasia. Clin Endocrinol (Oxf). 2013 May;78(5):667-72. doi: 10.1111/cen.12033. PMID 23057653
- [Background] Engels M, Span PN, van Herwaarden AE, Sweep FCGJ, Stikkelbroeck NMML, Claahsen-van der Grinten HL. Testicular Adrenal Rest Tumors: Current Insights on Prevalence, Characteristics, Origin, and Treatment. Endocr Rev. 2019 Aug 1;40(4):973-987. doi: 10.1210/er.2018-00258. PMID 30882882
- [Background] Al-Ghamdi WM, Shazly MA, Al-Agha AE. Testicular adrenal rest tumors in children with congenital adrenal hyperplasia. Saudi Med J. 2021 Sep;42(9):986-993. doi: 10.15537/smj.2021.42.9.20210257. PMID 34470837
- [Background] Chaudhari M, Johnson EK, DaJusta D, Nahata L. Testicular adrenal rest tumor screening and fertility counseling among males with congenital adrenal hyperplasia. J Pediatr Urol. 2018 Apr;14(2):155.e1-155.e6. doi: 10.1016/j.jpurol.2017.11.011. Epub 2017 Dec 21. PMID 29330018
- [Background] Eyer de Jesus L, Paz de Oliveira AP, Porto LC, Dekermacher S. Testicular adrenal rest tumors - Epidemiology, diagnosis and treatment. J Pediatr Urol. 2024 Feb;20(1):77-87. doi: 10.1016/j.jpurol.2023.10.005. Epub 2023 Oct 7. PMID 37845103
- [Background] Rivera-Hernandez A, Jimenez-Osorio M, Rodriguez-Mencias JP, Escamilla-Castaneda KM, Madrigal-Gonzalez MM, Zurita-Cruz J. Risk factors for testicular adrenal rest tumors in pediatric patients with congenital adrenal hyperplasia. J Pediatr Urol. 2023 Aug;19(4):398.e1-398.e7. doi: 10.1016/j.jpurol.2023.03.028. Epub 2023 Mar 24. PMID 37029011
- [Background] Stikkelbroeck NM, Otten BJ, Pasic A, Jager GJ, Sweep CG, Noordam K, Hermus AR. High prevalence of testicular adrenal rest tumors, impaired spermatogenesis, and Leydig cell failure in adolescent and adult males with congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2001 Dec;86(12):5721-8. doi: 10.1210/jcem.86.12.8090. PMID 11739428
- [Background] Tresoldi AS, Betella N, Hasenmajer V, Pozza C, Vena W, Fiamengo B, Negri L, Cappa M, Lania AGA, Lenzi A, Isidori AM, Pizzocaro A. Bilateral testicular masses and adrenal insufficiency: is congenital adrenal hyperplasia the only possible diagnosis? First two cases of TARTS described in Addison-only X-linked adrenoleukodystrophy and a brief review of literature. J Endocrinol Invest. 2021 Mar;44(3):391-402. doi: 10.1007/s40618-020-01362-x. Epub 2020 Jul 20. PMID 32691371